CLINICAL TRIAL: NCT04910373
Title: Determination of Hypoallergenicity of an Extensively Hydrolyzed Infant Formula in Infants and Children With Cow's Milk Allergy
Brief Title: Extensively Hydrolyzed Infant Formula in Infants and Children With Cow's Milk Allergy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Product Availability Due to Recall
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: AL36
Record Dates: First submitted 2021-05-18; First posted 2021-06-02 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Cow's Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Extensively Hydrolyzed Formula (Experimental): Administered during food challenge and at home feeding period
  Interventions: Other: Experimental Extensively Hydrolyzed Formula
- Placebo Extensively Hydrolyzed Formula (Placebo Comparator): Administered during food challenge
  Interventions: Other: Placebo Extensively Hydrolyzed Formula

INTERVENTIONS:
Other: Experimental Extensively Hydrolyzed Formula — experimental powder formula
  Arms: Experimental Extensively Hydrolyzed Formula
Other: Placebo Extensively Hydrolyzed Formula — placebo powder formula
  Arms: Placebo Extensively Hydrolyzed Formula

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled food challenge to be conducted in infants or children with confirmed IgE-mediated cow's milk allergy (CMA), followed by a 7-day open feeding of the experimental formula.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a physician diagnosis of IgE-mediated Cow's Milk Allergy (CMA) based on a clinical history of a reaction resulting in characteristic immediate hypersensitivity symptoms within 2 hours of oral exposure or immediate hypersensitivity symptoms according to physician's observation
* Participant is willing to undergo confirmatory testing or must have had at least one of the following within 6 months of enrollment:

  1. Documentation of milk-specific serum IgE >15 kIUA/L or > 5 kIUA/L if younger than 1 year.
  2. Documented cow's milk skin prick test mean wheal >10mm
  3. Physician-supervised oral food challenge that elicited immediate, objective, allergic symptoms.
* Participant agrees to stop oral steroid use within 14 days and antihistamine use within 7 days of confirmation of diagnosis and food challenges.
* Participant had followed a strict cow's milk protein-free diet prior to enrollment.
* Parent(s) confirm their intention not to administer any products containing cow's milk protein during the study.
* Participant's parent(s) has voluntarily signed and dated an Informed Consent Form (ICF), approved by an Independent Ethics Committee/Institutional Review Board (IEC/IRB) and provided Health Insurance Portability and Accountability Act (HIPAA) (or other applicable privacy regulation) authorization prior to any participation in the study.

Exclusion Criteria:

* Participant is exclusively breastfed at the time of enrollment.
* Participant is consuming an amino acid-based formula due to failure on an extensively hydrolyzed formula.
* Significant chronic medical diseases including major chromosomal or congenital anomalies, gastrointestinal diseases or abnormalities other than CMA, immunodeficiencies, unstable asthma, asthma treated with biologics (omalizumab or other monoclonal antibody), FPIES, eosinophilic esophagitis, and severe uncontrolled eczema.
* Previous severe anaphylactic reaction to cow's milk within the last two years.
* An adverse medical history or current condition that is thought by the investigator to have potential for effects on tolerance or the hypoallergenicity test.
* Participant has an allergy or intolerance to any ingredient in the study product, as reported by the parent.
* Participant is routinely consuming baked milk products.

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Food Challenge Positive Reactions | Food Challenge Day 1 to Food Challenge Day 2
  Percent of positive food challenge reactions to the experimental formula

SECONDARY OUTCOMES:
Experimental Formula Intake | Home Feeding Day 1 to Day 7
  Parent completed diaries of formula intake
Food Intake | Home Feeding Day 1 to Day 7
  Parent completed diaries
Gastrointestinal Symptoms | Home Feeding Day 1 to Day 7
  Parent completed diaries
Medication Use | Home Feeding Day 1 to Day 7
  Parent completed diaries
Food Challenge Positive Reactions | Home Feeding Day 1 to Day 7
  Percent of positive food challenge reactions to the experimental formula

CONTACTS AND LOCATIONS:
Overall Officials: Carlett Ramirez, Study Chair — Abbott Nutrition
Locations (4):
- United States (4):
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - UNC-Chapel Hill, Chapel Hill, North Carolina
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No